CLINICAL TRIAL: NCT04171193
Title: Efficacy of Deep Anaesthesia With Isoflurane as a Fast-response Antidepressant Agent in Treatment Resistant Depression Patients : Proof of Concept
Brief Title: Efficacy of Deep Anaesthesia With Isoflurane as a Fast-response Antidepressant Agent
Acronym: ISORADAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ricardo Alberto Moreno, M.D., Ph.D., DIRECTOR: MOOD DISORDERS UNIT (GRUDA), University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISORADAR; 19921719.9.0000.0068 (Other: Plataforma Brasil)
Record Dates: First submitted 2019-11-06; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Depressive Disorder, Major; Treatment Resistant Depression; Depressive Episode
Keywords: Isoflurane; Anesthesia; Treatment resistant depression; Deep anesthesia; Burst suppression; Depressive episode
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Isoflurane; Sertraline

STUDY DESIGN:
Intervention Model Description: We will have two groups, one arm with oral antidepressants and other arm without oral antidepressants, no placebo, no control. Everyone receives the intervention. Those who respond to treatment, will be followed for 24 weeks, those who do not respond, if not in the oral antidepressant group, will star oral antidepressants and be followed for 24 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ISO (Experimental): Patients not taking oral medications for depression. They will receive the study intervention consisting in general anesthesia with the volatile anesthetic gas Isoflurane until burst suppression is detected in electroencephalogram more than 80% of the time for 15 minutes.
  Interventions: Drug: Isoflurane
- ISOAD (Experimental): Patients in treatment with oral medications for depression, will receive intervention consisting in general anesthesia with the volatile anesthetic gas Isoflurane until burst suppression is detected in electroencephalogram more than 80% of the time for 15 minutes
  Interventions: Drug: Isoflurane
- ISOPOT (Experimental): Patients that where from ISO arm, that did not respond to intervention consisting in general anesthesia with the volatile anesthetic gas Isoflurane until burst suppression is detected in electroencephalogram more than 80% of the time for 15 minutes They will now, start taking sertraline as oral medication for depression to asset the enhancement of oral treatment after Isoflurane challenge.
  Interventions: Drug: Sertraline Pill

INTERVENTIONS:
Drug: Isoflurane — Deep anesthesia with isoflurane to achieve burst suppression pattern for more than 80% of the time for 15 minutes measured in electroencephalogram and Bi-Spectral Index
  Arms: ISO; ISOAD
Drug: Sertraline Pill — Patients that did not respond to Isoflurane treatment, will star on sertraline to evaluate any enhancement in antidepressant efficacy after pre-treatment with isoflurane
  Arms: ISOPOT

SUMMARY:
In this study the investigators will submit patients with treatment resistant depression to deep anesthesia with isoflurane to get 15 minutes of cortical burst suppression on electroencephalogram, once a week for six weeks. The follow up will be for 6 months. The aim is to evaluate the change in depression severity during the entire period.

DETAILED DESCRIPTION:
This study protocol will measure the efficacy of deep anesthesia, until burst suppression rate of 80% or more measured with Bi-spectral Index (BIS), with the volatile anesthetic Isoflurane. The investigators will select 30 subjects. The participants will be separated into 2 arms of 15 individuals. One arm called ISOAD will keep the oral treatment with antidepressants. The second arm, called ISO, will do a washout of any oral medications for depression. Both groups will go under six sessions, once per week, of deep anesthesia and will be followed up for 6 months to evaluate the survival of the antidepressant effect, if any effect happens. Before the anesthesia occurs, blood samples will be drawn to measure Brain-derived neurotrophic factor and investigators will apply depression rating scales such as MADRS and Hamilton - 17 , Young mania Scale, UKU scale for side effects, electroencephalogram will be recorder to be compared with the data shown on BIS. All the anesthesia procedure will be done with induction with propofol, fentanyl and muscular relaxant, to facilitate the tracheal intubation and compliance with the mechanical ventilator,based on body weight in standard dosages. Isoflurane will be set to 2,4% ( 2 cam) until Burst suppression rate >80% is achieve. Then the anesthesia will be maintained for 15 minutes, then the flow of anesthetic gas will be ended and the patient will be allowed to awake and discharged home when the anesthesiologist decide based on Aldrete Kroulik scale. After the 6th session the participant will return in one week to final evaluation. All the patients that shows improvement in depression scores will enter the phase 2 with one visit every 15 days for 2 months and then once a month until the 6th month. The non responders of the ISO group will start oral antidepressant sertraline to evaluate any potentialization effect of the intervention and be allocated in ISOPOT group. Those from ISOAD group (Isoflurane plus oral antidepressants) that did not respond to the intervention will be discontinued from the study and their data used in the study as non-responders. Those from ISOPOT group that did not improve their depression scores after 4 weeks will be discontinued from the study and the data computed as non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Treatment resistant depression on depressive state with or without psychiatric comorbidities for anxious features
* moderate to severe condition measured by Montgomery Asperger Depression Rating Scale and Hamilton Depression rating scale - 17
* be between 18 and 60 years old
* IF female, do not be pregnant and use a trustable contraceptive method
* can read and write in Portuguese language
* will to be in all the phases of the study
* have agreed with free will to participate
* classified as American Society of Anesthesiologists - Physical Status 1 or 2 by a certified anesthesiologist
* Suicide ideation measured by Montgomery Asperger Depression Rating Scale on item 10 less than 4

Exclusion Criteria:

* drug abusers in the last 6 months, except for nicotine
* use of benzodiazepines or lamotrigine less then 15 days from the first session
* family history of malignant hyperthermia Suicidal ideation on item 10 of Montgomery Asperger Depression Rating Scale more than 4
* Suicide attempt one month prior the study begins

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in Depression severity - MADRS | Six days after the last session
  Any reduction in Montgomery Asperger Depression Rating Scale ( 0 to 60 , lower score means less depression severity)
Reduction in Depression - HDRS 17 | Six days after the last session
  Any reduction in Hamilton Depression rating scale 17 ( 0 to 49, lower score means less depression severity

SECONDARY OUTCOMES:
Udvalg for Kliniske Undersøgelser - side effects rating scale | From 6th day after the first intervention up to week 24th
  Development and tolerability of collateral effects using the Udvalg for Kliniske Undersøgelser - side effects rating scale ( 0 to 43 - lower score means less side effects)
Change in Depression severity MADRS | From 6th day after the intervention up to week 24th
  Any change in Montgomery Asperger depression ratings scale ( 0 to 60 , lower score means less depression severity)
Change in Depression severity HDRS17 | From 6th day after the intervention up to week 24th
  Any change in Hamilton depression ratings scale 17 ( 0 to 49, lower score means less depression severity)
Magnitude MADRS | From 6th day after the intervention up to week 24th
  The amount of the reduction, if any, in Montgomery Asperger Depression Rating Scale ( 0 to 60 , lower score means less depression severity)
Magnitude HDRS 17 | From 6th day after the intervention up to week 24th
  The amount of the reduction, if any, in Hamilton Depression rating scale 17 ( 0 to 49, lower score means less depression severity)
Survival of the effect - HDRS 17 | After the 6th session through 24th week
  For how long the Hamilton Depression rating scale 17 remains below the initial value (lower value means less depression) in each participant that had variation in this scale
Survival of the effect - MADRS | After the 6th session through 24th week
  For how long the Montgomery Asperger Depression Rating Scale remains below the initial value (lower value means less depression) in each participant that had variation in this scale
Enhance HDRS 17 | After the 10th visit through the 24th week
  The magnitude, if any, of the change in Hamilton Depression rating scale 17 measured in patients that did not achieve any primary outcome in the first phase of the study after started sertraline as oral antidepressant.
Enhance MADRS | After the 10th visit through the 24th week
  The magnitude, if any, of the change in Montgomery Asperger Depression Rating Scale measured in patients that did not achieve any primary outcome in the first phase of the study after started sertraline as oral antidepressant.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Alberto Moreno, Phd, Study Director — Instituto de Psiquiatria do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Insitute of Psychiatry of the University of São Paulo, São Paulo, Brazil